CLINICAL TRIAL: NCT07331194
Title: A Single-Center, Open-Label, Randomized, Crossover Phase I Clinical Study to Evaluate the Pharmacokinetics and Bioequivalence of Two Different Formulations of HMPL-523 Acetate Tablets in Chinese Healthy Participants
Brief Title: Pharmacokinetics and Bioequivalence Study of HMPL-523 Acetate Tablets in Humans
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hutchmed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2025-523-00CH1
Record Dates: First submitted 2025-09-11; First posted 2026-01-09 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Healthy
Keywords: HMPL-523

STUDY DESIGN:
Intervention Model Description: Two formulations containing the same active pharmaceutical ingredient are considered bioequivalent if their relative bioavailability (rate and extent of drug absorption) falls within acceptable predetermined limits after administration at the same molar dose. Formulations with bioequivalence are considered to act comparably in vivo, i.e., similar in terms of safety and efficacy.
  This study aims to evaluate the pharmacokinetic (PK) profile and bioequivalence of the original and modified formulations of HMPL-523 acetate tablets in healthy participants to bridge the safety and efficacy of the modified formulation of HMPL 523 acetate tablets in humans.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TRTR (Other): Total 54 Chinese healthy participants are planned to be enrolled and randomly assigned to 2 dosing sequence groups (TRTR, and RTRT) in a 1:1 ratio and administered once per cycle, with a washout period of at least 7 days, where T is the test formulation (the modified formulation) and R is the reference formulation (the original formulation). the dose is 300mg for each cycle, and there were 4 cycles for each participant.
  Interventions: Drug: HMPL-523 Acetate Tablets (Test Formulation); Drug: HMPL-523 Acetate Tablets (Reference Formulation)
- RTRT (Other): Total 54 Chinese healthy participants are planned to be enrolled and randomly assigned to 2 dosing sequence groups (TRTR, and RTRT) in a 1:1 ratio and administered once per cycle, with a washout period of at least 7 days, where T is the test formulation (the modified formulation) and R is the reference formulation (the original formulation). the dose is 300mg for each cycle, and there were 4 cycles for each participant.
  Interventions: Drug: HMPL-523 Acetate Tablets (Test Formulation); Drug: HMPL-523 Acetate Tablets (Reference Formulation)

INTERVENTIONS:
Drug: HMPL-523 Acetate Tablets (Test Formulation) — The trial participants were administered the drug on the first day of each cycle. dose 300mg
Drug: HMPL-523 Acetate Tablets (Reference Formulation) — The trial participants were administered the drug on the first day of each cycle. dose 300mg

SUMMARY:
Two formulations containing the same active pharmaceutical ingredient are considered bioequivalent if their relative bioavailability (rate and extent of drug absorption) falls within acceptable predetermined limits after administration at the same molar dose. Formulations with bioequivalence are considered to act comparably in vivo, i.e., similar in terms of safety and efficacy.

This study aims to evaluate the pharmacokinetic (PK) profile and bioequivalence of the original and modified formulations of HMPL-523 acetate tablets in healthy participants to bridge the safety and efficacy of the modified formulation of HMPL 523 acetate tablets in humans.

DETAILED DESCRIPTION:
This study adopts a single-center, randomized, open-label, single-dose, four-cycle, fully replicate clinical trial design to evaluate the PK profile and bioequivalence of two different formulations of HMPL-523 acetate tablets in healthy participants. In this study, a total of 54 Chinese healthy participants are planned to be enrolled and randomly assigned to 2 dosing sequence groups (TRTR, and RTRT) in a 1:1 ratio, and administered once per cycle, with a washout period of at least 7 days, where T is the test formulation (the modified formulation) and R is the reference formulation (the original formulation).

The study will be divided into 3 periods: screening/baseline period, dosing period (four cycles), and follow-up period. The entire study from the screening period to the follow-up period is expected to last approximately 2 months.

Screening Period/Baseline Period The trial participants will sign a written informed consent form (ICF) on a voluntary basis prior to screening. Screening period/baseline period assessment will be completed within 14 days prior to the first dose. At screening/baseline, demographic data, medical history, medication history, allergy history, blood donation history, and participation in clinical trials should be collected, and physical examination, vital sign measurements, alcohol breath test, urine drug abuse screening, 12-lead ECG, infection markers [including hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antibody, and Treponema pallidum antibody], laboratory tests (including hematology, blood chemistry, coagulation test, urinalysis), pregnancy test (female) and chest X-ray (frontal and lateral) examination will be performed. Only serious adverse events (SAEs) will be collected at screening/baseline.

Dosing Period (4 cycles) Eligible participants upon preliminary screening will be required to be admitted to the site 3 days before the first dose (i.e., 3 days prior to the initiation of the first cycle of medication). On the day of admission, vital sign measurements and inquiry about recent diet and medication, and pregnancy test (females only) will be performed to further verify the inclusion and exclusion criteria. According to the randomization scheme, eligible participants upon screening will be assigned a random number and randomly assigned to different dosing sequences (TRTR or RTRT). Based on the randomized dosing regimen, participants in different groups will take the test formulation or the reference formulation respectively after intake of breakfast (standard meal) on the first day of each cycle. The dosing regimen is detailed in the table below.

Crossover dosing regimen Group Number of participants Intake of standard meal breakfast Cycle 1 Cycle 2 Cycle 3 Cycle 4 TRTR 27 T R T R RTRT 27 R T R T

Method of administration:

Participants will fast for at least 10 hours before a standard meal on the first day of each cycle, start having a standard meal 30 minutes before dosing, and finish the meal within 25 minutes. After the meal, participants will have blank blood samples collected, and take the medication with about 240 mL of water on time 30 minutes after the meal. Except for the above-mentioned water for medication, participants are deprived of water is prohibited from 1 hour prior to the medication to 1 hour after the medication, and deprived of food within 4 hours after the medication. During hospitalization, the diet of the participants will be provided by the site.

The dosing period consists of four cycles, and the scheduled PK blood sampling time points for each participant in each cycle is as follows: within 0.5 hours pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 12, 24, 36, 48, 60, 72 hours post-dose, with a total of 18 collections (see Table 2 for details), and about 3 mL of venous blood collected each time.

After the participants are admitted to the clinical study ward, the vital sign measurements will be performed 1 day pre-dose in each cycle and 3±1 hours post-dose on the first day of each cycle. In addition, vital sign measurements, blood chemistry, and hematology will be performed on the Day 4 of the each of the first three cycles. On Cycle 4 Day 4, the participants will be discharged after vital sign measurements, physical examination, laboratory tests, and 12-lead ECG examination are completed.

Follow-up Period Participants will be followed up to Day 12±2 after the last dose (the day of the last dose is defined as Day 1 of follow-up period). The investigator will collect all AEs and concomitant medications/therapies from the participants during this period through telephone calls (or other means such as text messages). If there are AEs ongoing at follow-up, follow-up will continue until return to normal level, abnormal, not clinically significant, baseline level, stable or lost to follow-up, or refusal to visit, etc.,

ELIGIBILITY:
Inclusion Criteria:

Trial participants must meet all of the following criteria for enrollment:

1. Participants can communicate well with the investigator, must voluntarily sign the ICF and agree to comply with the requirements of the study protocol;
2. Male and female healthy participants aged 18-45 years (inclusive);
3. Body weight ≥ 45 kg (females) or ≥ 50 kg (males), body mass index (BMI) 19-26 kg/m2 (inclusive);
4. Study participants must commit to using highly effective contraception for both themselves and their sexual partners during the study, and for 180 days after the end of the last study dose, and must not engage in sperm donation, egg donation, or have birth plan.

Exclusion Criteria:

Study participants must be excluded from this study if one of the following conditions is met:

1. Abnormal and clinically significant results of vital signs, physical examination, 12-lead ECG, chest X-ray (frontal and lateral), laboratory tests (including hematology, blood chemistry, urinalysis, etc.) or serum creatinine above the upper limit of normal at screening;
2. Positive for any of the HBsAg, HCV antibody, HIV antibody, or Treponema pallidum antibody;
3. History or current evidence of severe or chronic metabolic/endocrine, hepatic, renal, hematological, pulmonary, immunological, cardiovascular, gastrointestinal, genitourinary, neurological or psychiatric diseases;
4. Prior history of hypertension;
5. Prior history of severe gastrointestinal diseases such as dysphagia, active gastric ulcers, etc., resulting in inability to take oral medication or disorders in absorption of oral medication
6. Prior history of gastrointestinal surgery, renal surgery, cholecystectomy, etc. that, in the judgment of the investigator, may affect drug absorption or excretion;
7. Prior history of drug allergy, or acute allergic rhinitis or food allergy within 2 weeks before screening, or allergy to the active ingredients or excipients of the study drug;
8. Use of any prescription drugs and Chinese herbal medicines within 30 days prior to the first dose;
9. Use of any over-the-counter drugs, vitamins, and health products within 14 days prior to the first dose;
10. Consumption of more than 10 cigarettes per day within 3 months before screening, or those who cannot quit smoking during the study;
11. Regular alcohol consumption within 6 months before screening, that is, those who drink more than 14 units of alcohol per week (1 unit = 360 mL of beer, or 45 mL of spirits with an alcohol content of 40%, or 150 mL of wine), or those who cannot abstain from alcohol during the study, or those who are positive for alcohol breath test;
12. History of drug abuse or recreational use, or positive for urine drug abuse screen;
13. Blood donation (including blood component donation) or blood loss ≥ 400 mL within 3 months prior to screening, blood products within 2 months prior to screening, blood donation (including component blood donation) or lost blood ≥ 200 mL within 1 month prior to screening, or a plan to donate blood or blood components during the study or within 1 month after the end of the study;
14. Difficulty in blood collection, or a history of needle phobia or blood phobia, or intolerance to blood sampling via venipuncture, or poor evaluation of venous blood collection;
15. Participants who participated in clinical studies of other drugs/medical devices and received investigational drugs within 3 months prior to screening;
16. Participants who have consumed foods, juices or drinks containing alcohol, grapefruit, Seville oranges and caffeine within 72 hours before the first dose, or cannot avoid them during the study;
17. Those who have received live vaccines within 8 weeks prior to screening or have plans to vaccinate during the clinical study;
18. Those who have special requirements for diet and cannot accept unified dietary arrangements;
19. Pregnant or lactating women, or those with blood pregnancy test results above the upper limit of normal during screening, or women with unprotected sex within 2 weeks prior to dosing;
20. The study participant, based on the judgment of the investigator, has any other diseases or conditions that may affect the normal completion of the study or the evaluation of study data, or other conditions that make him/her unsuitable for participation in this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2025-10-28 (Actual); Primary Completion 2025-11-28 (Actual); Study Completion 2026-02-02 (Actual)

PRIMARY OUTCOMES:
PK parameters | up to two months
  area under the plasma concentration-time curve from 0 to the time point t when the last concentration can be accurately measured (AUC0-t)
PK parameters | up to two months
  area under the plasma concentration-time curve from 0 to infinity (AUC0-∞)
PK parameters | up to two months
  maximum concentration (Cmax)
PK parameters | up to two months
  time to maximum concentration (Tmax)
PK parameters | up to two months
  terminal elimination half-life (t1/2)
The bioequivalence of two different drug product formulations of HMPL 523 acetate tablets | up to two months
  It will be evaluated based on the area under the plasma concentration-time curve (AUC) and Cmax.

SECONDARY OUTCOMES:
To compare the relative bioavailability of two different drug product formulations of 300 mg (100 mg/tablet × 3) HMPL-523 acetate tablets | up to two months
  Relative bioavailability (ratio of AUC of two different HMPL-523 acetate tablets)
Adverse events (AEs) | up to two months
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
Laboratory tests | up to two months
  Number of participants with abnormal laboratory tests results

CONTACTS AND LOCATIONS:
Overall Officials: Bin Yang, Study Director — Hutchmed
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University, Jinan, Shandong, China